CLINICAL TRIAL: NCT00139386
Title: Effects of Candesartan Cilexetil on Cardiovascular Events in Japanese Patients With Hypertension After Sirolimus- or Paclitaxel-Eluting Stents Implantation
Brief Title: Candesartan for Prevention of Cardiovascular Events After Cypher or Taxus Coronary Stenting (4C) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Collaborators: The 4C trial bureau (Unknown); Japan Heart Foundation (Other)
Responsible Party: Principal Investigator, Hisao Ogawa, MD, PhD, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVM-RCT-2005-01
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension; Coronary Artery Disease
Keywords: Drug-eluting stent; Candesartan; Randomized control study; Coronary Angioplasty
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Candesratan (Active Comparator)
  Interventions: Drug: Candesartan
- Non-candesartan (No Intervention)

INTERVENTIONS:
Drug: Candesartan — Candesartan Cilexetil (4-12 mg per day)
  Other Names: Blopress; 4C
  Arms: Candesratan

SUMMARY:
Candesartan is effective in preventing cardiovascular events in patients without restenosis after coronary angioplasty. Therefore, the investigators hypothesized that candesartan after drug-eluting stent (DES) implantation was also effective in preventing cardiovascular events.

The purpose of this study is to investigate whether an angiotensin II receptor blocker, candesartan, is effective in reducing the incidence of cardiovascular events after drug-eluting stent implantation.

DETAILED DESCRIPTION:
It was reported that low-dose angiotensin II receptor blocker, candesartan, was effective to prevent cardiovascular events in patients with coronary artery disease treated with coronary angioplasty (Am Heart J 146:E20, 2003). In this study, patients without significant coronary stenosis on follow-up angiography 6 months after intervention were randomly assigned into a candesartan group (baseline treatment plus candesartan 4 mg/d) or a control group (baseline treatment alone). It is well known that patients treated with drug-eluting stents (DES) have lower restenosis rate as compared with those with bare metal stents. Therefore, we hypothesized that candesartan started immediately after DES implantation was effective to prevent cardiovascular events.

The primary endpoint is a composite of any cause death and cardiovascular events (nonfatal myocardial infarction, recurrent symptomatic myocardial ischemia, congestive heart failure, and stroke). The secondary endpoints are target lesion revascularization, binary restenosis, newly onset diabetes and newly onset of atrial fibrillation.

Patient population which needs to prove the hypothesis is estimates to be 1,130 cases in total (565 cases in each group). We set the parameters which are needed to calculate the number of study patients as follows; a drop out rate 10%, an event rate of the primary end point for 3 years 20%, a risk reduction rate brought by candesartan 25%, a statistical power 90% and a two-sided significance level 0.05. We assumed the event rate from the study which was conducted to prove the effects of statins after PCI in Japan named MUSASHI-PCI. Also the risk reduction rate from two major RCTs of candesartan conducted in Japan named the Ogaki and HIJ-CREATE studies. In the Ogaki study, the risk reduction rate by candesartan was 52%. However, stents used in the study were only BMS after surviving restenosis. The risk reduction of the present study will be lower because of the higher onset rate of stent thrombosis in regard to DES. Furthermore, the risk reduction rate of candesartan for Japanese was 11% reported in HIJ-CREATE. The ACE-I usage rate was almost 70% in the control subjects of HIJ-CREATE. In the present study, ACE-I will be administered less frequently as low as 30%. Therefore, assumed risk reduction rate by candesartan in the present study could be higher. Considering all the various factors together, a reasonable risk reduction rate could be 25%.

ELIGIBILITY:
Inclusion Criteria:

* A. Patients with hypertension, systolic blood pressure (SBP) = or > 140 and/or diastolic blood pressure (DBP) = or > 90
* B. Patients with symptomatic heart failure lasting at least for 4 weeks (NYHA class = or > II), or those need continuous use of diuretics
* C. Patients underwent coronary angioplasty with drug-eluting stents

Eligible patients are those who meet (A or B) and C.

Exclusion Criteria:

* Severe renal or hepatic disease
* Candidates for coronary artery bypass grafting (CABG)
* Within 3 months after CABG
* Allergic history to candesartan
* Pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1119 (Actual)
Dates: Start 2005-10; Primary Completion 2009-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite of: 1)any cause mortality and 2)cardiovascular events (non-fatal MI, drug-resistant AP required hospital admission, heart failure required hospital admission and stroke) | 3 years

SECONDARY OUTCOMES:
Target lesion revascularization | 3 years
Binary restenosis | 3 years
Newly onset diabetes | 3 years
Newly onset atrial fibrillation | 3 yeard
Each of the primary endpoint events | 3 years
  All cause of death, cardiovascular death, non-fatal myocardial infarction, unstable angina required admission, heart failure required admission and stroke
Major adverse cardiac-related events | 3 years
  A composite of cardiovascular death, non-fatal myocardial infarction, unstable angina required admission and heart failure required admission
Major cardiac-related events | 3 years
  A composite of non-fatal myocardial infarction, unstable angina required admission and heart failure required admission

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University
Locations (1):
- Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University, Kumamoto, Japan

REFERENCES:
- [Background] Kondo J, Sone T, Tsuboi H, Mukawa H, Morishima I, Uesugi M, Kono T, Kosaka T, Yoshida T, Numaguchi Y, Matsui H, Murohara T, Okumura K. Effects of low-dose angiotensin II receptor blocker candesartan on cardiovascular events in patients with coronary artery disease. Am Heart J. 2003 Dec;146(6):E20. doi: 10.1016/S0002-8703(03)00443-5. PMID 14661009
- [Derived] Sakamoto T, Ogawa H, Nakao K, Hokimoto S, Tsujita K, Koide S, Yamamoto N, Shimomura H, Matsumura T, Oshima S, Kikuta K, Oka H, Kimura K, Matsui K; 4C (Candesartan for Prevention of Cardiovascular Events after CYPHER or TAXUS Coronary Stenting) study investigators. Impact of candesartan on cardiovascular events after drug-eluting stent implantation in patients with coronary artery disease: The 4C trial. J Cardiol. 2016 Apr;67(4):371-7. doi: 10.1016/j.jjcc.2015.06.009. Epub 2015 Aug 4. PMID 26254019
- See also: Dept of CVM, Kumamoto Univ Hosp — http://www.kumadai-junnai.com/